CLINICAL TRIAL: NCT07138612
Title: The Effect of Peer Education in Urinary Catheterization on Students' Skill Levels, Privacy Awareness, Anxiety and Satisfaction Levels
Brief Title: The Effect of Peer Education in Urinary Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Asst. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TarsusU-NBARISEREN-006
Record Dates: First submitted 2025-08-16; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Nursing Education
Keywords: peer education; nursing education; nursing student

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Education Group (Experimental): Five peer educators will be randomly selected from among students who agree to participate in the study. Peer education will be provided 2 weeks before the implementation date. After students are randomly assigned to experimental and control groups, the experimental group will be divided into five subgroups. Each group consists of seven students. A peer educator will be assigned to lead each group. Before the implementation, students will complete the Sudent Information Form, the Urinary Catheterization Checklist, the Privacy Awareness Scale, and the State Anxiety Inventory (STAI-I). Peer educators will work with students in groups on a mock-up during the practical part of the theoretical course. The topic will be reinforced using a well-equipped mock-up. All students will complete the Urinary Catheterization Checklist, the Privacy Awareness Scale, and the State Anxiety Inventory (STAI-I) as a post-test. Additionally, students in the intervention group will complete the "Satisfaction
  Interventions: Behavioral: Peer education group
- Control Group (No Intervention): Students will be randomly assigned to an experimental and control group, and then the control group will be divided into five subgroups. Each group will consist of seven students. Before the intervention, students will complete the Sudent Information Form, the Urinary Catheterization Checklist, the Privacy Awareness Inventory, and the State Anxiety Inventory (STAI-I). No intervention will be made. Students in the control group will receive their education in the traditional manner. The topic will be reinforced using a rigged mannequin. All students will take the Urinary Catheterization Checklist, the Privacy Awareness Inventory, and the State Anxiety Inventory (STAI-I) as a posttest. To assess the retention of learning, the Urinary Catheterization Checklist will be administered one week later as a posttest.

INTERVENTIONS:
Behavioral: Peer education group — Students will learn urinary catheterization through peer education.
  Arms: Peer Education Group

SUMMARY:
This study aimed to evaluate the effects of peer education in urinary catheterization on students' skill levels, privacy awareness, anxiety, and satisfaction levels.

Hypotheses:

H1. Peer education in urinary catheterization increases students' skill levels. H2. Peer education in urinary catheterization increases students' privacy awareness.

H3. Peer education in urinary catheterization reduces students' anxiety levels. H4. Peer education in urinary catheterization increases students' satisfaction levels.

DETAILED DESCRIPTION:
This study evaluated the effects of peer education on urinary catheterization on students' skill levels, privacy awareness, anxiety, and satisfaction. It was found that peer education increased students' urinary catheterization skills and privacy awareness, reduced anxiety levels, and enhanced satisfaction levels. Based on these results, it was suggested that using peer education in the teaching of other nursing practices could also increase nursing students' privacy awareness, reduce anxiety levels, and improve satisfaction levels. This educational method, particularly in a critically important nursing practice course, was expected to enhance students' knowledge and skills and improve learning retention. Furthermore, peer education made learning more enjoyable, which was anticipated to increase student engagement, motivation, and satisfaction. This study revealed a significant difference in how nursing students, and future nurses, interacted with patients and their families. This difference contributed to improved quality of patient care and positively affected patient and family satisfaction. Additionally, receiving positive feedback after nursing practices carried out with confidentiality awareness was found to increase employee satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being 18 years of age or older
* Being a first year student
* Taking the Fundamentals of Nursing course for the first time
* Not being a student who came via horizontal or vertical transfer
* Not having received training on 'Urinary Catheterization'
* Not having been absent on the dates when the research data will be collected

Exclusion Criteria:

* Not volunteering to participate in the research
* Being under 18 years old
* Not being a first year student
* Being a student who came via horizontal or vertical transfer

  -- Having received training on 'Urinary Catheterization'
* Being a health vocational high school graduate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Student Information Form | 10 minutes
  It was prepared by the researcher by scanning the relevant literature and consists of 14 questions regarding the sociodemographic characteristics, personal information and peer education of the students participating in the study.
Urinary Catheterization Checklist | 20 minutes
  This checklist was created by researchers with expertise in the field of nursing fundamentals (Göçmen Baykara et al., 2021). The "Urinary Catheterization Checklist" is a checklist systematically designed to evaluate urinary catheterization. The checklist is a 3-point Likert-type scale with markings of "incompletely implemented," "fully implemented," or "not implemented." Students will receive 2 points for fully implementing the practice step, 1 point for incomplete implementation, and 0 points for not implementing. No feedback will be given to students while administering the checklists to assess their skill levels. Feedback will be provided following the evaluation. All student evaluations will be conducted by the same instructor.
Privacy Awareness Scale | 10 minutes
  It was developed by Tabata and Sato (2014) to measure privacy awareness in nursing students. The validity and reliability study of the scale in the Turkish language was conducted by Öztürk et al. (2019). Each item is a 5-point Likert-type scale with a score between 1 and 5. 1 represents "strongly disagree," 2 represents "disagree," 3 represents "undecided," 4 represents "agree," and 5 represents "strongly agree." The scale includes three subfactors: privacy awareness of oneself/behaviors to maintain privacy of self (4 items: 2, 4, 6, 10), privacy awareness for others (4 items: 1, 5, 8, 11), and behaviors to maintain privacy of others (3 items: 3, 7, 9), and contains a total of 11 items. The scale contains eight reverse-scored items (2, 4, 6, 10, 1, 5, 3, and 7). For each subscale, the scores from the items representing the subscale are summed, and the means are compared to evaluate the total score. The highest possible score is 55, and the lowest is 11. However, when the mean scores a
State Anxiety Inventory (STAI-I) | 10 minutes
  The State Anxiety Inventory (STAI-I) was developed by Spielberger and colleagues (1970). It was adapted into Turkish by Öner and Le Compte (1998). The scale consists of 20 questions and measures how an individual feels at a specific moment and under a specific circumstance. The response options on the state anxiety scale are categorized into four classes: (1) Not at all, (2) A little, (3) A lot, and (4) Completely. The scale contains ten reversed statements: items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The fixed value for the State Anxiety Inventory is 50. The state anxiety score is obtained by subtracting the total score for reversed statements from the total score for direct statements and adding the predetermined fixed value. The fixed value for the State Anxiety Scale is 50. Theoretically, scores obtained on the State Anxiety Scale range from 20 to 80. In the evaluation of the scale, scores below 36 are considered to indicate no anxiety, between 37 and 42 to indicate mild anxiety
Satisfaction Assessment with Peer Education | 10 minutes
  Students who received peer education were asked to give a score between 1 and 10 to determine their level of satisfaction with the education after the research. 1- not at all, 10- very much, and they were asked to give a full score.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No